CLINICAL TRIAL: NCT03131869
Title: Development of Novel, Biophysically Designed Fluids for Swallowing Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Swallow Solutions (Industry)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2R44NR015193-02 (NIH); 2R44NR015193-02 (NIH)
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Deglutition Disorders
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Thickened Beverages Nectar — Thickened beverages in nectar consistency
Other: Thickened Beverage Honey — Thickened beverages in honey consistency

SUMMARY:
People suffering from swallowing disorders (dysphagia) have a hard time swallowing liquids that are too thin (like water or coffee) or too thick, correctly. They can have health problems, such as chest infections and malnutrition because when they try to drink, some of the liquid "goes down the wrong pipe" and into the lungs. To help people with dysphagia, Swallow Solutions is developing thickened liquids that have added nutrition, taste good, and quench thirst, but are still easy and safe to swallow.

DETAILED DESCRIPTION:
A. Background Dysphagia, a devastating swallowing disorder affecting more than 18M adults and millions more children in the U.S. [1,2], is associated with increased mortality and morbidity, including malnutrition, dehydration, pulmonary complications, and reduced quality of life [3,4]. Dysphagia often causes thin liquids (e.g., water, coffee) to be aspirated or misdirected into the pulmonary-rather than to the digestive-system during swallowing, significantly increasing the risk of aspiration pneumonia [5,6]. Radiographic methods used in >80% of U.S. hospitals to diagnose dysphagia involve standardized fluids with specific rheological characteristics (e.g., apparent viscosity, flow properties) [7]. Thickened beverages are the most commonly recommended intervention after dysphagia diagnosis [8]. Perplexingly, currently available dietary beverages differ from the rheological characteristics of standardized diagnostic fluids, causing a critical disconnect between diagnosis and treatment [9]. A rheologic study of commercially available thickened beverages and diagnostic fluids found that some commercial nectar products, while approaching the target apparent viscosity (n ) for the diagnostic standard (Varibar® Nectar, n 30=300 cP), differed in other rheological parameters such as flow index (n), consistency (K), and yield stress. o commercial thin-honey consistency products matched the diagnostic standard for any of these rheological parameters. This disconnect frequently causes the bolus to flow toward the airway, increasing the risk of negative health sequelae.

Swallow Solutions, LLC will build on the successful completion of our Phase I project to continue to bridge the gap between clinical need and existing products. Based on insights from our Phase I results, investigators will develop a complete product line (tentatively branded as SwallowSAFE Thickened Beverages) to meet the unique-currently unmet-needs of dysphagic patients. This novel thickened beverage line will provide hydration and nutrition, thus circumventing potentially life-threatening and costly health problems associated with dysphagia. The investigators propose to accomplish the following specific aims.

Specific Aims

Aim 1. Complete a full complement of prototype ready-to-drink, thickened, and nutritionally-enhanced medical liquids that are shelf-stable and appealing, with pre-determined rheological and nutritional properties. T

Aim 2. Demonstrate improved patient safety resulting from novel, biophysically designed thickened beverages (full product line) compared to currently available thickened beverage options.

Aim 3. Develop production for the full SwallowSAFE product line of ready-to-drink, thickened beverages (with and without nutritional enrichment) at 2 target viscosities (nectar and thin-honey) in 1-3 flavors each.

B. Study Design: Clinical Research (Aim 2)

Dysphagic patients (n=200) will swallow prototype beverages (with 10% added barium) and also thickened beverages that are currently on the market (with 10% added barium) during a videofluoroscopic (radiographic) evaluation of swallowing that is part of their standard clinical care. The investigators will use established, quantified, objective safety measures of a) airway invasion (Penetration/Aspiration Scale) [13,14] and b) oropharyngeal residue [15]. Potential subjects will be adults (age >55 years) with suspected dysphagia based on referral for the diagnostic evaluation. The study will include patients with a variety of medical etiologies to allow for greater generalizability of results. Each consenting subject will complete a videofluoroscopic swallowing assessment lasting ~45 min per standard clinical care. Data will be collected from 200 subjects from two large acute-care hospitals.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* physician approval of medical stability
* aspiration or penetration of the laryngeal vestibule (score of 3 or higher on the Penetration/Aspiration Scale) or post-swallow residue in the oropharynx as instrumentally documented by a Speech-Language Pathologist (SLP) during a standard videofluoroscopic oropharyngeal swallow study
* capacity to provide informed consent.

Exclusion Criteria:

* poorly controlled psychosis (3 or more related hospitalizations in one year
* refractory alcoholism (on AWD precautions)
* allergy to barium (used in radiographic swallowing assessment)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects will be adults with suspected dysphagia based on referral for a diagnostic videofluoroscopic swallowing evaluation. Only subjects who can consent for themselves will be enrolled in the study. The consent will take place before the swallow study begins. The study will include patients with a variety of medical etiologies to allow for greater generalizability of results. Pregnant women will be excluded from this protocol. Per standard clinical care (as all subjects will be completing the radiologic procedure regardless of participation in the study), pregnancy test will not be required.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-02-22 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Penetration - Aspiration Scale | immediately while swallowing
  presence of aspiration/penetration of the laryngeal vestibule

SECONDARY OUTCOMES:
Post-swallow Residue | immediately while swallowing
  quantification of oropharyngeal residue

CONTACTS AND LOCATIONS:
Overall Officials: Eric Horler, MBA, Principal Investigator — Swallow Solutions; JoAnne Robbins, PhD, Principal Investigator — Swallow Solutions
Locations (2):
- United States (2):
  - Meriter Hospital, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No